CLINICAL TRIAL: NCT00717782
Title: Randomized Clinical Trial of Botulinum Toxin Injection for Pain Relief in Patients With Thrombosed External Haemorrhoids
Brief Title: Pain Relief for Thrombosed External Haemorrhoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Gaetano Di Vita, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIPA001
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Thrombosed External Hemorrhoid
Keywords: botulinum toxin; thrombosed external haemorrhoids; pain
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients were injected with 0·6 ml of a solution containing 30 units botulinum toxin A (Botox; Allergan, Ireland).
  A 27-G needle was used to give two injections of equal volume (0·3 ml) into the internal anal sphincter, one on each side of the anterior midline of the sphincter.
  Interventions: Procedure: injection of botulinum toxin
- 2 (Placebo Comparator): Patients in the placebo group received a 0·6-ml injection of saline.
  A27-G needle was used to give two injections of equal volume (0·3 ml) into the internal anal sphincter, one on each side of the anterior midline of the sphincter.
  Interventions: Procedure: injection of saline

INTERVENTIONS:
Procedure: injection of botulinum toxin — Patients received a 0·6-ml injection of a solution containing 30 units botulinum toxin into the internal anal sphincter
  Other Names: botox injection
  Arms: 1
Procedure: injection of saline — Patients received a 0·6-ml injection of a saline solution into the internal anal sphincter
  Other Names: saline injection
  Arms: 2

SUMMARY:
Thrombosed external haemorrhoids are one of the most frequent anorectal emergencies. They are associated with swelling and intense pain. This study evaluated the efficacy and safety of an intersphincteric injection of botulinum toxin for pain relief in patients with thrombosed external haemorrhoids

DETAILED DESCRIPTION:
Background: Thrombosed external haemorrhoids are one of the most frequent anorectal emergencies. They are associated with swelling and intense pain. Internal sphincter hypertonicity plays a role in the aetiology of the pain. This study evaluated the efficacy and safety of an intersphincteric injection of botulinum toxin for pain relief in patients with thrombosed external haemorrhoids. Methods: Thirty patients with thrombosed external haemorrhoids who refused surgical operation were randomized into two groups. Patients received an intrasphincteric injection of either 0·6 ml saline or 0·6 ml of a solution containing 30 units botulinum toxin. Anorectal manometry was performed before treatment and 5 days afterwards.Results: After 5 days of treatment, the maximum resting pressure fell in both groups, but was significantly lower in the botulinum toxin group (P = 0·004). Pain intensity was significantly reduced within 24 h of botulinum toxin treatment (P < 0·001), but only after 1 week in the placebo group (P = 0·019). Conclusion: A single injection of botulinum toxin into the anal sphincter seems to be effective in rapidly controlling the pain associated with thrombosed external haemorrhoids, and could represent an effective conservative treatment for this •condition.

ELIGIBILITY:
Inclusion Criteria:

* thrombosed external haemorrhoids disease
* patients that refused surgery for fear of procedure related pain.

Exclusion Criteria :

* previous anal surgery
* third- and fourth-degree haemorrhoids
* anal fissure
* anal fistula
* presumed or confirmed pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy and safety of intrasphincteric injection of botulinum toxin for pain relief in patients with Thrombosed External Haemorrhoids. | 1

SECONDARY OUTCOMES:
evaluate the absence of side-effects and the simplicity of application | 1

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Di Vita, Principal Investigator — A.O.U.P.; Rosalia Patti, Study Chair — A.O.U.P.

REFERENCES:
- [Derived] Patti R, Arcara M, Bonventre S, Sammartano S, Sparacello M, Vitello G, Di Vita G. Randomized clinical trial of botulinum toxin injection for pain relief in patients with thrombosed external haemorrhoids. Br J Surg. 2008 Nov;95(11):1339-43. doi: 10.1002/bjs.6236. PMID 18844269